CLINICAL TRIAL: NCT05817318
Title: Renal Denervation in Patients With Recurrent Atrial Fibrillation After Successful Pulmonary Vein Isolation (REDE-AF): a National, Multi-centre, Prospective, Single-arm, Pre-to-post Treatment, Medical-device Study
Brief Title: Renal Denervation in Patients With Recurrent Atrial Fibrillation After Successful Pulmonary Vein Isolation
Acronym: REDE-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REDE-AF
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Arrhythmia Burden in Patients With Recurrent, Paroxysmal Atrial Fibrillation Despite Durable Pulmonary Vein Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-to-post renal denervation treatment (Other): Pre-to-post treatment comparison
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation — Arrhythmia burden pre-to-post renal denervation as assessed by an implantable cardiac monitor

SUMMARY:
The aim of this study is to investigate whether renal denervation can reduce arrhythmia burden in patients with recurrent, paroxysmal atrial fibrillation despite durable pulmonary vein isolation.

DETAILED DESCRIPTION:
Pulmonary vein isolation is the treatment of choice in symptomatic patients with paroxysmal atrial fibrillation. Despite durable pulmonary vein isolation, 15% of patients continue to have episodes of atrial fibrillation because of triggers of atrial fibrillation localized outside the pulmonary veins. Additional ablation of these triggers is difficult because they often cannot be localized. The autonomous nervous system does influence these triggers and modulation of the autonomous nervous system with the goal to reduce sympathetic activity may be an alternative approach to suppress these extra-pulmonary vein triggers. Renal denervation does reduce sympathetic activity and is successfully used to treat drug-resistant arterial hypertension. The combination of pulmonary vein isolation with renal denervation has already been shown to be superior to pulmonary vein isolation alone in patients with paroxysmal atrial fibrillation regarding arrhythmia-free outcome. The investigators hypothesize that renal denervation can suppress atrial fibrillation in patients with recurrent episodes of paroxysmal atrial fibrillation despite durable isolation of the pulmonary veins.

The best way to assess atrial fibrillation burden is with an implantable cardiac monitor (ICM), which the investigators will use both before and after renal denervation, to gather detailed data on daily atrial fibrillation burden.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* ≥ 18 years of age
* Recurrent, paroxysmal atrial fibrillation post repeat (≥2) pulmonary vein isolation
* Documentation of atrial fibrillation ≥3 months after the last atrial fibrillation ablation procedure by a 12-lead ECG or on a rhythm strip of ≥30 seconds duration
* Either an office systolic blood pressure ≥130 mmHg at the screening visit or antihypertensive drug therapy

Exclusion Criteria:

* Persistent or permanent atrial fibrillation post pulmonary vein isolation
* Left ventricular ejection fraction <40%
* Severe aortic or mitral valve stenosis
* Treatment with amiodaron within the last 3 months
* Mandatory treatment with class I or III antiarrhythmic drugs
* History of reflex syncope, syncope due to orthostatic hypotension or unclear syncope in the past 3 years.
* History of orthostatic hypotension
* Abnormal blood pressure fall during active standing, defined as a progressive and sustained fall in systolic blood pressure from baseline value ≥20 mmHg or diastolic blood pressure ≥10mmHg, or a decrease in systolic blood pressure to <90 mmHg.
* Prior renal denervation
* Renal artery stent or prior renal angioplasty
* Polycystic kidney disease, unilateral kidney, or history of renal transplant
* Estimated glomerular filtration rate (eGFR) < 50mL/min, using the CKD-EPI creatinine equation (Chronic Kidney Disease Epidemiology)
* Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy.
* Life expectancy <1 year
* Enrolment in interventional studies if the other study does not allow enrolment or if primary endpoint might be affected by study participation.
* Diabetes mellitus type I
* Aortic grafts

The following exclusion criteria will apply after the run-in phase of up to 3 months duration, prospectively in patients which receive a new ICM and retrospectively in patients which already have an ICM implanted:

- Episodes of atrial fibrillation on <6 days in the 3 months run-in phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in atrial fibrillation burden | 6 months
  The primary endpoint is the atrial fibrillation burden in the 6 months following renal denervation compared to the 3 months before renal denervation as assessed by the ICM.

SECONDARY OUTCOMES:
Freedom from atrial fibrillation recurrence | 12 months
  Freedom from atrial fibrillation recurrence at 12 months after renal denervation
Time to first atrial fibrillation recurrence after renal denervation | 12 month
Change in mean number of days with atrial fibrillation | 6 months
  Mean number of days with atrial fibrillation in the 6 months following renal denervation compared to the 3 months before, as assessed by the ICM.
Evolution of AF burden measured as mean number of days with atrial fibrillation in the 12 months following renal denervation, as compared to before renal denervation | 12 months
  Evolution of AF burden measured as mean number of days with atrial fibrillation in the 12 months following renal denervation, as compared to before renal denervation
Evolution of AF burden measured as mean number of days with atrial fibrillation in the 3 years following renal denervation, as compared to before renal denervation | 3 years
  Evolution of AF burden measured as mean number of days with atrial fibrillation in the 3 years following renal denervation, as compared to before renal denervation
Change in arterial blood pressure after renal denervation | 3 months
  Arterial blood pressure 3 months after renal denervation compared to before (24-hours ambulatory blood pressure measurements).
Change in arterial blood pressure after renal denervation | 12 months
  Arterial blood pressure 12 months after renal denervation compared to before (24-hours ambulatory blood pressure measurements).
Change in day heart rate following renal denervation | 12 months
  Day heart rate following renal denervation compared to before, as assessed by the ICM.
Change in patient activity | 12 months
  Patient activity following renal denervation compared to before, as assessed by the ICM
Change in heart rate variability | 12 months
  Heart rate variability following renal denervation compared to before, as assessed by the ICM.
Change in arterial blood pressure after renal denervation | 3 months
  Arterial blood pressure 3 months after renal denervation compared to before (office blood pressure measurements).
Change in arterial blood pressure after renal denervation | 12 month
  Arterial blood pressure 12 months after renal denervation compared to before (office blood pressure measurements).
Change in night heart rate following renal denervation | 12 months
  Night heart rate following renal denervation compared to before, as assessed by the ICM.

OTHER OUTCOMES:
Blood pressure | 12 months
  Abnormal blood pressure fall during active standing, defined as a progressive and sustained fall in systolic blood pressure from baseline value ≥20 mmHg or diastolic blood pressure
  ≥10mmHg, or a decrease in systolic blood pressure to <90 mmHg
Procedure-related complications of renal denervation | 12 hours
  Renal artery perforation or dissection requiring intervention
Procedure-related complications of renal denervation | 1 month
  Vascular complications (e.g., clinically significant groin hematoma, arteriovenous fistula, pseudoaneurysm, excessive bleeding, or distal microembolization causing visible circulatory impairment to the lower limbs) requiring surgical repair, interventional procedure, thrombin injection, or blood transfusion.
Renal artery perforation or dissection requiring intervention | 1 year
  New renal artery stenosis > 70%, confirmed by angiography

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Roten, Prof, Principal Investigator — Insel Gruppe AG
Locations (2):
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern

IPD SHARING:
Plan to Share IPD: No